CLINICAL TRIAL: NCT02250209
Title: Trastuzumab Plus XELOX for HER2-positive Stage III Gastric Cancer After D2 Gastrectomy：Prospective Observational Study.
Brief Title: T- XELOX in HER2-positive Stage III Gastric Cancer After D2 Gastrectomy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Dai, Guanghai, Professor and chief physician, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGOG20130101005
Record Dates: First submitted 2014-09-24; First posted 2014-09-26 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; HER2-positive; Trastuzumab; XELOX; Stage III; D2 Gastrectomy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Trastuzumab; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trastuzumab,Capecitabine,Oxaliplatin (Experimental): Patients receive eight 3-week cycles of oral capecitabine (800-1000 mg/m2 twice daily on days 1-14 of each cycle) ,intravenous oxaliplatin (130 mg/m2 on day 1 of each cycle) plus intravenous Trastuzumab (440mg on day 0 of each cycle).
  Number of cycle:capecitabine and oxaliplatin --8 cycles; Trastuzumab--14-16 cycles.
  Interventions: Drug: Trastuzumab; Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab is given by intravenous infusion at 440mg on day 0every 3 weeks. Number of cycles: 14~16 cycles.
  Other Names: Herceptin; Herclon
Drug: Capecitabine — Capecitabine 800~1000 mg/m² is given orally twice a day for 14 days followed by a 1-week rest.
  Number of cycles: 8 cycles.
  Other Names: Xeloda
Drug: Oxaliplatin — Oxaliplatin is given by intravenous infusion at 130 mg/m2 on day 1 every 3 weeks.
  Number of cycles: 8 cycles.
  Other Names: Eloxatin

SUMMARY:
The objective of this study is to assess the clinical efficacy and safety of trastuzumab plus XELOX for treatment of HER2-positive Stage III Gastric Cancer After D2 Gastrectomy.

DETAILED DESCRIPTION:
Gastric cancer is the second leading cause of cancer death worldwide. Highest incidence rate is observed in Eastern Asia.

D2 gastrectomy has been established as a standard surgical procedure. While recurrence rate after resection is still high.

The CLASSIC study showed that Xelox regimen after D2 gastrectomy improves 3-year disease-free survival compared with surgery only. But patients with late stage still have poor prognosis according to subgroup analysis and our retrospective study.

HER2 is an important biomarker and key driver of tumorigenesis in 7-34% gastric cancers. The ToGA study showed that trastuzumab, a monoclonal antibody that targets HER2, plus chemotherapy improved overall survival(16.0m vs 11.8m) in patients with HER2-positive advanced gastric or gastro-oesophageal junction cancer.

Based on previous experiences of trastuzumab in adjunctive therapy of breast cancer and ACTS/CLASSIC/ToGA studies, we suppose that trastuzumab plus XELOX as adjunctive treatment may benefit patients with HER2-positive Stage III gastric cancer after D2 Gastrectomy.

According to the above, we do this single-arm research to assess the clinical efficacy and safety of trastuzumab plus XELOX for treatment of HER2-positive Stage III Gastric Cancer After D2 Gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed-consent form.
2. Aged 18-80 years.
3. Had partial or total D2 gastrectomy and achieved R0 resection.
4. Histologically confirmed gastric or gastro-oesophageal junction adenocarcinoma，mucinous adenocarcinoma ，signet-ring cell carcinoma
5. Pathologic Stage III (IIIA-C).
6. HER2-positive: (IHC 3+ or IHC 2+ and FISH positive).
7. Patients must have received no preoperative chemotherapy or radiation therapy.
8. Eastern Cooperative Oncology Group (ECOG) performance status 0-2 .
9. Adequate liver/bone marrow function.Blood and biochemical parameters;
10. Compliant, and can be followed up regularly.

Exclusion Criteria:

1. Patients who do not meet the Inclusion Criteria.
2. Pregnant or breast-feeding female, or not willing to take contraception measures during study.
3. Serious infection requiring antibiotics intervention during recruitment.
4. Allergic to study drug or with metabolism disorder.
5. Histologically confirmed small cell carcinoma of the stomach、gastric neuroendocrine carcinoma or others.
6. Uncontrolled brain metastasis or mental illness.
7. Organ transplant recipients (Autologous transplantation of bone marrow and peripheral stem cell transplantation included).
8. Congestive heart failure, uncontrolled cardiac arrhythmia, etc.
9. With severe hepatic/kidney/respirator/disease,or chronic disease like uncontrolled diabetes,hypertension,etc.
10. with other malignant tumors.
11. Can be followed up or obey protocol.
12. Ineligible by the discretion of the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival (DFS) | Measure at every 6 weeks (every 2 cycles)
  Defined as the time from study treatment to the time of recurrence of the original gastric cancer, development of a new gastric cancer, or death from any cause.

SECONDARY OUTCOMES:
Overall survival | up to 3 years
  Measure of time from study treatment to patient's death or lost to follow-up.
Safety and tolerability | up to 18 month
  Percentage of patients who experience adverse events during this study.
Prognostic value of biomarkers | up to 3 years
  assessment of the relationship between biomarker status and prognosis

CONTACTS AND LOCATIONS:
Overall Officials: Guanghai Dai, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Bang YJ, Kim YW, Yang HK, Chung HC, Park YK, Lee KH, Lee KW, Kim YH, Noh SI, Cho JY, Mok YJ, Kim YH, Ji J, Yeh TS, Button P, Sirzen F, Noh SH; CLASSIC trial investigators. Adjuvant capecitabine and oxaliplatin for gastric cancer after D2 gastrectomy (CLASSIC): a phase 3 open-label, randomised controlled trial. Lancet. 2012 Jan 28;379(9813):315-21. doi: 10.1016/S0140-6736(11)61873-4. Epub 2012 Jan 7. PMID 22226517
- [Result] Gravalos C, Jimeno A. HER2 in gastric cancer: a new prognostic factor and a novel therapeutic target. Ann Oncol. 2008 Sep;19(9):1523-9. doi: 10.1093/annonc/mdn169. Epub 2008 Apr 25. PMID 18441328
- [Result] Hofmann M, Stoss O, Shi D, Buttner R, van de Vijver M, Kim W, Ochiai A, Ruschoff J, Henkel T. Assessment of a HER2 scoring system for gastric cancer: results from a validation study. Histopathology. 2008 Jun;52(7):797-805. doi: 10.1111/j.1365-2559.2008.03028.x. Epub 2008 Apr 18. PMID 18422971
- [Result] Tanner M, Hollmen M, Junttila TT, Kapanen AI, Tommola S, Soini Y, Helin H, Salo J, Joensuu H, Sihvo E, Elenius K, Isola J. Amplification of HER-2 in gastric carcinoma: association with Topoisomerase IIalpha gene amplification, intestinal type, poor prognosis and sensitivity to trastuzumab. Ann Oncol. 2005 Feb;16(2):273-8. doi: 10.1093/annonc/mdi064. PMID 15668283
- [Result] Piccart-Gebhart MJ, Procter M, Leyland-Jones B, Goldhirsch A, Untch M, Smith I, Gianni L, Baselga J, Bell R, Jackisch C, Cameron D, Dowsett M, Barrios CH, Steger G, Huang CS, Andersson M, Inbar M, Lichinitser M, Lang I, Nitz U, Iwata H, Thomssen C, Lohrisch C, Suter TM, Ruschoff J, Suto T, Greatorex V, Ward C, Straehle C, McFadden E, Dolci MS, Gelber RD; Herceptin Adjuvant (HERA) Trial Study Team. Trastuzumab after adjuvant chemotherapy in HER2-positive breast cancer. N Engl J Med. 2005 Oct 20;353(16):1659-72. doi: 10.1056/NEJMoa052306. PMID 16236737
- [Result] Slamon DJ, Leyland-Jones B, Shak S, Fuchs H, Paton V, Bajamonde A, Fleming T, Eiermann W, Wolter J, Pegram M, Baselga J, Norton L. Use of chemotherapy plus a monoclonal antibody against HER2 for metastatic breast cancer that overexpresses HER2. N Engl J Med. 2001 Mar 15;344(11):783-92. doi: 10.1056/NEJM200103153441101. PMID 11248153
- [Result] Bang YJ, Van Cutsem E, Feyereislova A, Chung HC, Shen L, Sawaki A, Lordick F, Ohtsu A, Omuro Y, Satoh T, Aprile G, Kulikov E, Hill J, Lehle M, Ruschoff J, Kang YK; ToGA Trial Investigators. Trastuzumab in combination with chemotherapy versus chemotherapy alone for treatment of HER2-positive advanced gastric or gastro-oesophageal junction cancer (ToGA): a phase 3, open-label, randomised controlled trial. Lancet. 2010 Aug 28;376(9742):687-97. doi: 10.1016/S0140-6736(10)61121-X. Epub 2010 Aug 19. PMID 20728210
- [Result] Smith I, Procter M, Gelber RD, Guillaume S, Feyereislova A, Dowsett M, Goldhirsch A, Untch M, Mariani G, Baselga J, Kaufmann M, Cameron D, Bell R, Bergh J, Coleman R, Wardley A, Harbeck N, Lopez RI, Mallmann P, Gelmon K, Wilcken N, Wist E, Sanchez Rovira P, Piccart-Gebhart MJ; HERA study team. 2-year follow-up of trastuzumab after adjuvant chemotherapy in HER2-positive breast cancer: a randomised controlled trial. Lancet. 2007 Jan 6;369(9555):29-36. doi: 10.1016/S0140-6736(07)60028-2. PMID 17208639
- [Result] Dai GH, Shi Y, Chen L, Lv YL, Zhong M. Trastuzumab combined with docetaxel-based regimens in previously treated metastatic gastric cancer patients with HER2 over-expression. Hepatogastroenterology. 2012 Nov-Dec;59(120):2439-44. doi: 10.5754/hge12166. PMID 22534547
- [Result] Terashima M, Kitada K, Ochiai A, Ichikawa W, Kurahashi I, Sakuramoto S, Katai H, Sano T, Imamura H, Sasako M; ACTS-GC Group. Impact of expression of human epidermal growth factor receptors EGFR and ERBB2 on survival in stage II/III gastric cancer. Clin Cancer Res. 2012 Nov 1;18(21):5992-6000. doi: 10.1158/1078-0432.CCR-12-1318. Epub 2012 Sep 12. PMID 22977193
- [Result] Okines AF, Thompson LC, Cunningham D, Wotherspoon A, Reis-Filho JS, Langley RE, Waddell TS, Noor D, Eltahir Z, Wong R, Stenning S. Effect of HER2 on prognosis and benefit from peri-operative chemotherapy in early oesophago-gastric adenocarcinoma in the MAGIC trial. Ann Oncol. 2013 May;24(5):1253-61. doi: 10.1093/annonc/mds622. Epub 2012 Dec 11. PMID 23233651
- [Result] Sasako M, Sakuramoto S, Katai H, Kinoshita T, Furukawa H, Yamaguchi T, Nashimoto A, Fujii M, Nakajima T, Ohashi Y. Five-year outcomes of a randomized phase III trial comparing adjuvant chemotherapy with S-1 versus surgery alone in stage II or III gastric cancer. J Clin Oncol. 2011 Nov 20;29(33):4387-93. doi: 10.1200/JCO.2011.36.5908. Epub 2011 Oct 17. PMID 22010012